CLINICAL TRIAL: NCT06264167
Title: Randomised Feasibility Study of Groin Ultrasound Surveillance to De-Escalate Surgical Intervention in Queensland Women With Vulvar Cancer
Brief Title: NODE (groiN ultrasOunD cancEr)
Acronym: NODE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queensland Centre for Gynaecological Cancer (Other Government)
Collaborators: Royal Brisbane and Women's Hospital (Other Government); St Andrew's War Memorial Hospital (Other); Buderim Private Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NODE
Record Dates: First submitted 2024-01-09; First posted 2024-02-16 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Vulvar Cancer Stage Ib; Vulvar Cancer Stage II; Lymph Node Metastasis; Groin Node; Ultrasound Therapy; Complications
Keywords: Vulvar Cancer; Ultrasound Therapy
MeSH Terms: conditions — Vulvar Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Intervention Model Description: Feasibility trial, open label, three-group, randomised clinical trial
  30 eligible females aged 18 or older with clinically stage 1b or 2 vulvar cancer will receive a bilateral groin node ultrasound up to 30 days prior to planned surgery:
  Participants with normal/negative baseline groin ultrasounds will be randomly assigned to two groups (2:1 randomisation): one group undergoing radical procedures (groin lymph nodes are not removed) with bilateral groin ultrasound surveillance in conjunction with clinical examinations every 2 months, and the other group undergoing upfront full groin LND or sentinel node biopsy (SNB) based on clinician choice (according to local clinical practice management guidelines).
  Participants with suspicious/indeterminate baseline groin ultrasound (third group) will receive an upfront full groin LND or SNB, consistent with the current standard treatment, according to local clinical practice management guidelines.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Participants with normal/negative baseline groin ultrasounds (Experimental): Interventional Treatment: serial high-resolution bilateral groin ultrasound surveillance in conjunction with clinical examinations every 2 months (n=13).
  Interventions: Diagnostic Test: High-resolution bilateral groin ultrasound surveillance
- Participants with normal/negative baseline groin ultrasounds - Standard Care (No Intervention): Standard Treatment: receive upfront full groin LND or sentinel node biopsy (SNB) based on clinician choice (according to local clinical practice management guidelines).
- Participants with suspicious/indeterminate baseline groin ultrasound (No Intervention): Participants with suspicious/indeterminate baseline groin ultrasound (third group) will receive an upfront full groin LND or SNB, consistent with the current standard treatment, according to local clinical practice management guidelines.

INTERVENTIONS:
Diagnostic Test: High-resolution bilateral groin ultrasound surveillance — Participants in the Interventional Treatment (serial ultrasounds) group will undergo surgical excision of the primary tumor, either via radical wide local excision or radical vulvectomy. Post-vulvar surgery, follow-up appointments occur bi-monthly for 12 months, involving a clinical examination and groin ultrasound. Senior imaging specialists review bilateral ultrasound scans for positive lymph nodes or suspicious findings, promptly sending reports to the primary care physician and trial manager if detected within 3 business days. Subsequently, participants consult their primary care physician for options. Depending on clinical judgment, they may be referred for LND or continue with bi-monthly ultrasounds based on preference and clinician guidance.
  Arms: Participants with normal/negative baseline groin ultrasounds

SUMMARY:
This study is an open label, prospective, experimental, randomised clinical trial. The primary aim of this study is to determine whether it is feasible to randomise vulvar cancer patients into one of two treatment arms:1) surgical groin node dissection (as delivered though either a sentinel node biopsy or inguinofemoral lymph node dissection (IFL), or 2) serial high-resolution bilateral groin ultrasound surveillance and clinical examination every 2 months.

DETAILED DESCRIPTION:
Treatment of vulvar cancer causes significant morbidity. Despite being a rare cancer, at least 2500 survivors of vulvar cancer live in Australia. Most survivors live with the detrimental, life-long impacts resulting from their cancer treatment because there are currently no alternatives to mitigate these impacts. The personal and societal burden this entails is significant. To control such cancer-associated burden is a national priority.

Clinical palpation of the groin region and computed tomography (CT) scans do not reliably detect groin node involvement. Hence, current clinical guidelines recommend all women diagnosed at apparent Stage I or II have a surgical groin LND. This can be performed as a full IFL (full LND) to remove all groin nodes, or as a SNB to remove selected (one or two) nodes. SNB is less invasive, however, is appropriate only for vulvar cancers <4cm in diameter and unifocal tumours (~50% of all Stage I and II vulvar cancers). SNB is also associated with a false negative rate (10%) that increases the risk of undetected nodes.

In 25% of cases (~80 Australian women per year), groin LND will reveal positive nodes (i.e., metastases), which triggers a referral for radiation treatment. If positive groin nodes are missed, and over time become enlarged, clinically palpable and attached to the overlying skin, >90% of women will die within 12 months, despite subsequent treatment. Conversely, if groin node involvement is detected early (e.g., by ultrasound) while still small, survival outcomes are excellent. Ultrasound technology is potentially as accurate as LND due to recent advances in resolution and technologies such as 2D/3D volumetric assessments and tissue flow. Furthermore, ultrasound is superior to medical resonance imaging (MRI), and to standard CT and positron emission tomography (PET) scans in capturing groin node involvement because it has a higher resolution, avoids harmful radiation and the technology is readily accessible outside of high-volume metropolitan areas.

The investigators propose to reduce surgical morbidity by replacing upfront groin LND for vulvar cancer patients with serial high-resolution ultrasound to detect groin metastases. Groin LND will only be necessary for the few women with ultrasound-detected metastases when they are still small. This feasibility study (NODE - groiN ultrasOunD cancer) will determine the value of randomized serial groin ultrasound examinations in stage I and II vulvar cancer patients and whether it is feasible and safe for the investigators to de-escalate the extent of vulvar cancer surgery, aiming to achieve improved outcomes for affected patients.

Australian women with this rare cancer bear an unacceptably high (and potentially avoidable) treatment-related burden. This feasibility study is the first step to address this problem in a novel yet pragmatic way. The overall outcome of NODE is a novel, less invasive alternative to vulvar cancer LND associated with significantly less morbidity, without compromising survival.

ELIGIBILITY:
Inclusion Criteria:

* Women, over 18 years, with histologically confirmed SCC, adenocarcinoma or melanoma of the vulva
* Clinically stage I or II on medical imaging (CT scan of pelvis, abdomen, and chest), without evidence of regional or distant metastatic disease
* Participant must be suitable to undergo IFL/SNB according to local clinical practice management guidelines
* Signed written informed consent
* Negative serum pregnancy test ≤ 30 days of surgery in pre-menopausal women and women < 2 years after the onset of menopause
* Patient lives within 40 km of a medical diagnostic imaging centre (site investigator approval required for special circumstances)

Exclusion Criteria:

* Women with non-invasive vulvar conditions (e.g. non-invasive non-mammary Paget's disease)
* Squamous cell carcinoma (SCC) of the vulva with depth of invasion ≤1 mm
* Clinical or medical imaging evidence of regional and/or distant metastatic disease
* Serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator)
* Other prior malignancies <5 years before inclusion, except for successfully treated keratinocyte skin cancers, or ductal carcinoma in situ
* Estimated life expectancy of ≤6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of randomisation: The percentage of patients willing to be randomised to either surgical groin node dissection or serial high-resolution bilateral groin ultrasound surveillance in conjunction with clinical examination every 2 months. | 12 months
  The feasibility of randomisation into (1) LND (IFL vs SNB) or (2) high-resolution bilateral groin ultrasound surveillance every 2 months will be determined through a practical sample size of n=20. Feasibility is declared if 30% of eligible patients (n=6 or more) can be randomised.

SECONDARY OUTCOMES:
Utility of tumour mutations to determine positive lymph node metastasis. | Study duration up to 15 years
  Translational research - Compare the molecular profile of tumour mutations between positive and negative lymph nodes.
Utility of circulating tumour DNA to determine positive lymph node metastasis. | Study duration up to 15 years
  Translational research - Compare the molecular profile of circulating tumour DNA between positive and negative lymph nodes.
Utility of plasma to determine positive lymph node metastasis. | Study duration up to 15 years
  Translational research - Compare the molecular profile of plasma between positive and negative lymph nodes.
Utility of serum to determine positive lymph node metastasis. | Study duration up to 15 years
  Translational research - Compare the molecular profile of serum between positive and negative lymph nodes.

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - St Andrew's War Memorial Hospital, Brisbane, Queensland
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Buderim Private Hospital, Sunshine Coast, Queensland

IPD SHARING:
Plan to Share IPD: No